CLINICAL TRIAL: NCT01185366
Title: Everolimus Versus Sunitinib Therapy in Patients With Advanced Non-clear Cell Renal Cell Carcinoma
Brief Title: Everolimus Versus Sunitinib in Non-Clear Cell Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0628; NCI-2012-01789 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Kidney Cancer
Keywords: Advanced non-clear cell renal cell cancer (RCC); Clear-cell renal cell carcinoma; Collecting duct carcinoma; Translocation carcinoma; Chromophobe; Everolimus; Sunitinib; Afinitor; RAD001; Sunitinib Malate; SUO11248; Sutent; ESPN
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Everolimus; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Everolimus Group 1 (Experimental): Everolimus 10 mg by mouth once a day.
  Interventions: Drug: Everolimus
- Sunitinib Group 2 (Active Comparator): Sunitinib 50 mg by mouth daily for 4 weeks on / 2 weeks off.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Everolimus — 10 mg by mouth once a day.
  Other Names: Afinitor; RAD001
  Arms: Everolimus Group 1
Drug: Sunitinib — 50 mg by mouth daily for 4 weeks on / 2 weeks off
  Other Names: Sunitinib Malate; SUO11248; Sutent
  Arms: Sunitinib Group 2

SUMMARY:
The goal of this clinical research study is to compare the effectiveness of Afinitor (everolimus) and Sutent (sunitinib) for the treatment of advanced renal cell carcinoma (kidney cancer). The safety of each treatment will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Everolimus is designed to stop cells from multiplying. It may also stop the growth of new blood vessels that help tumor growth, which may cause the tumor cells to die.

Sunitinib is designed to block pathways that control important events (such as the growth of blood vessels) that are essential for the growth of cancer.

Study Groups and Study Drug Administration:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups.

* If you are assigned to Group 1, you will take 2 everolimus tablets by mouth once every day.
* If you are assigned to Group 2, you will take sunitinib capsules by mouth every day for 4 weeks, followed by 2 weeks off.

If you have any side effects from any of the drugs, tell the study doctor right away. The study doctor may then lower the dose or keep the dose level the same.

Every 6 weeks on this study is called a study "cycle."

If the disease gets worse or you have intolerable side effects while you are on study, you will have the chance to receive the study drug that you did not receive at first. The dosing and follow-up will be the same as for all participants in that group.

Study Visits:

On Day 1 of every cycle:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any drugs or treatments you may be receiving.
* Your performance status will be recorded.
* Blood (about 3 teaspoons) and urine will be collected for routine tests and a fasting blood sugar test. Blood or urine will also be used for a pregnancy test for women who are able to have children. If you are in Group 1, you will have an additional 1 teaspoon of blood drawn to test your cholesterol.

On Day 15 and 29 of Cycle 1:

* Your vital signs and weight will be measured.
* Blood (about 2 teaspoons) will be drawn for routine tests. If you are in Group 1, an additional 1 teaspoon of blood will be drawn to measure your cholesterol.

The Day 15 and Day 29 tests may be done at your local doctor's office.

On Day 1 of Cycles 2 and 3, and every other cycle after that (Day 1 of Cycle 5, 7, 9 and so on):

°You will have a CT scan of the chest and a CT scan or MRI of the abdomen to check the status of the disease.

Every 4 cycles (24 weeks):

°If you are in Group 2, you will have an echocardiogram or MUGA scan to check your heart's health.

Length of Study:

You may continue taking the study drugs for as long as you are benefiting. You will be taken off study if the disease gets worse or intolerable side effects occur.

End-of-Treatment Visit:

If you have stopped taking the study drug because of intolerable side effects, the treating physician will make every effort to check the status of the disease before you are taken off of study.

Long-Term Follow-up:

Once you are no longer on this study, the research staff will check up on you about every 6 months. This update will consist of a phone call or a review of your medical and/or other records. You will not have any extra tests, procedures, or study visits. If contacted by phone, the call would only last about 5 minutes.

This is an investigational study. Sunitinib and everolimus are both FDA approved and commercially available for the treatment of advanced kidney cancer.

Up to 108 patients will be enrolled in this multicenter trial. Up to 108 patients will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have advanced non-clear cell RCC, which may include but is not limited to the following subtypes: papillary I or II, chromophobe, collecting duct carcinoma (CDC), translocation or unclassified. Patients with conventional-type renal cell carcinoma who have >/= 20% sarcomatoid component in their primary tumor are eligible. Patients who have sarcomatoid features in FNA or core biopsy of any metastatic site are eligible, if they have an underlying renal cell carcinoma primary tumor.
2. Patients must have at least one measurable site of disease that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation
3. ECOG performance status 0-1
4. Age >/= 18 years
5. Patients must have adequate organ and marrow function within 14 days prior to study entry as defined below: a) Hemoglobin >/= 9 g/dl (tx allowed); b) absolute neutrophil count >/=1,500/microL; c) platelets >/= 100,000/microL; d) total bilirubin </= 1.5 mg/dl; e) AST(SGOT) or ALT (SGPT) </=2.5 X institutional uln, except in known hepatic metastasis, wherein may be </= 5 x ULN; f) Serum Creatinine </= 1.5 x ULN (as long as patient does not require dialysis)
6. INR and PTT </= 1.5 x ULN within 14 days prior to study entry. Therapeutic anticoagulation with warfarin is allowed if target INR </= 3 on a stable dose of warfarin or on a stable dose of LMW heparin for > 2 weeks (14 days) at time of randomization.
7. Fasting serum cholesterol </= 300 mg/dL OR </= 7.75 mmol/L AND fasting triglycerides </= 2.5 x ULN within 14 days prior to study entry.
8. Female patients of childbearing potential (not postmenopausal for at least 12 months and not surgically sterile) must have a negative serum or urine pregnancy test within 14 days before study entry. Pregnancy test must be repeated if performed > 14 days before starting study drug.
9. Patients must give written informed consent prior to study entry, in keeping with the policies of each institution.
10. Patients with a history of major psychiatric illness must be judged (by the treating physician) able to fully understand the investigational nature of the study and the risks associated with the therapy.
11. Patients with controlled brain metastases are allowed on protocol if they had solitary brain metastases that was surgically resected or treated with radiosurgery or Gamma knife, without recurrence or edema for 3 months (90days).

Exclusion Criteria:

1. No other malignancies within the past 2 years except for adequately treated carcinoma of the cervix or basal (without recurrence post-surgery or post-radiotherapy) or squamous cell carcinomas of the skin.
2. No prior systemic therapy for RCC including prior adjuvant therapy or investigational drug is allowed.
3. Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks (28 days) from enrollment into this study (including chemotherapy and targeted therapy) are excluded. However, patients are permitted to receive bisphosphonates. Also, patients who completed palliative radiation therapy prior to enrollment in this trial are eligible.
4. Patients, who have had a major surgery or significant traumatic injury (injury requiring > 4 weeks (28 days) to heal) within 4 weeks (28 days) of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study.
5. Concomitant treatment with rifampin, St. John's wort, or the cytochrome p450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or Phenobarbital) or CYP3A4 inhibitors is not recommended on this study.
6. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: a) Symptomatic congestive heart failure of New York heart Association Class III or IV; b) unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease; c) severely impaired lung function as defined as 02 saturation that is 88% or less at rest on room air
7. (#6 cont'd) d) uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN; e) active (acute or chronic) or uncontrolled severe infections requiring antibiotic intervention; f) liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
8. Patients must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of sunitinib or everolimus or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
9. Concomitant treatment with drugs with dysrhythmic potential (terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, and indapamide) is not recommended.
10. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
11. Patients should not receive immunization with attenuated live vaccines within one week (7 days) of study entry or during study period.
12. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
13. A known history of HIV sero-positivity.
14. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus and/or sunitinib (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
15. Patients with an active, bleeding diathesis.
16. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to study entry. Pregnancy test must be repeated if performed > 7 days before administration of everolimus and sunitinib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amado Zurita, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Dana-Farber Cancer Institute/Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute - University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 73 Participants recruited from August 2010 to November 2013 at MD Anderson and Dana-Farber/Harvard Cancer Center.
Pre-assignment Details: 73 participants were recruited, 1 Screen failure. 69 participants were evaluable. Eligible patients did not take systemic medication for advanced papillary, chromophobe, CDC, Xp11.2 translocation, unclassified RCC or ccRCC with ≥ 20% sarcomatoid features in their primary tumors.
Groups:
- Everolimus: 4 weeks of everolimus of 10 mg orally each day then 2 weeks of no medication until progression. At progression will crossover to sunitinib.
- Sunitinib: 4 weeks of sunitinib of 50 mg orally each day then 2 weeks of no medication until progression. At progression will crossover to everolimus.
Period: First Line Therapy
Arm/Group | Everolimus | Sunitinib
Started | 38 | 34
Received 1st Drug | 36 | 33
Completed | 35 | 33
Not Completed | 3 | 1
Not completed — Insurance Coverage Denied | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lack of Metastatic Site | 1 | 0
Period: Crossover to Second Line Therapy
Arm/Group | Everolimus | Sunitinib
Started | 35 | 33
Received Crossover Drug | 21 | 23
Completed | 21 | 23
Not Completed | 14 | 10
Not completed — Adverse Event | 3 | 6
Not completed — Physician Decision | 5 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Continued with 1st drug | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus | Sunitinib | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Continuous [Median (Full Range); unit: years] | 58 [23 to 73] | 60 [28 to 76] | 60 [23 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 24 | 19 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 29 | 25 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 28 | 25 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 05 | 5 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 33 | 68
Histology [Count of Participants; unit: Participants] — Pathology description of baseline biopsy
  Participants
    Papillary | 13 | 14 | 27
    Clear Cell with sarcomatoid features | 6 | 6 | 12
    Chromophobe | 6 | 6 | 12
    Translocation | 4 | 3 | 7
    Unclassified | 6 | 4 | 10
ECOG Performance Score [Number; unit: participants] — Participants baseline ability for self-care, activity and physical ability: score 0-5. 0 is fully active. 1 is light house work and office work. 2 is cannot carry out work activities but up and about 50% of waking hours. 3 is limited to bed or chair more than 50% of waking hours 4. Completely disabled. 5. Dead
  participants
    0 | 15 | 18 | 33
    1 | 20 | 15 | 35
    2 | 0 | 0 | 0
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0
    5 | 0 | 0 | 0
Memorial Sloan Kettering Risk Group [Number; unit: participants] — Score based on participants performance score, time from diagnosis to treatment, hemoglobin count, lactate dehydrogenase level, and corrected calcium levels. O score is a good prognosis. 1 -2 is an intermediate prognosis, 3-5 is a poor prognosis
  participants
    Good | 4 | 4 | 8
    Intermediate | 29 | 29 | 58
    Poor | 2 | 0 | 2
International Metastatic RCC Database Consortium Risk Score for Renal Cell Carcinoma (RCC) [Number; unit: participants] — Score based on participant's time from diagnosis to treatment, performance score, hemoglobin counts calcium level, neutrophil count, and platelet count. 0 is a good risk. 1-2 is an intermediate risk. 3-5 is a poor risk.
  participants
    Good | 4 | 3 | 7
    Intermediate | 24 | 26 | 50
    Poor | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) for First Line Medication
Description: The amount of time after the first line medication begins until the cancer gets worse progresses. Progression is measured by an increase in measures tumors of at least 20 %, or overall increase in all the tumors, or the presence of new tumors.
Time Frame: 7 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus | Sunitinib
Number analyzed (Participants) | 35 | 33
months | 4.1 [2.7 to 10.5] | 6.1 [4.2 to 9.4]

2. Primary Outcome: Progression Free Survival (PFS) for Crossover Medication
Description: The amount of time after the crossover medication begins until the cancer gets worse progresses. Progression is measured by an increase in measures tumors of at least 20 %, or overall increase in all the tumors, or the presence of new tumors.
Time Frame: 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus | Sunitinib
Number analyzed (Participants) | 21 | 23
months | 1.8 [1.4 to 10.6] | 1.8 [1.4 to NA] — insufficient number of participants with events

3. Secondary Outcome: Number of Participants Who Experienced Either a Grade 3 or 4 Adverse Event
Description: Side effects, also called adverse events, that were related to either drug were documented and graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3. Grades increases in severity from 1 - 5. Grade one is a mild change which only requires monitoring. Grade 2 is a moderate change and may require some medication. Grade 3 is severe and requires hospitalization. Grade 4 is life threatening. Grade 5 is death.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Everolimus: 4 weeks of everolimus of 10 mg orally each day then 2 weeks of no medication until progression.
- Sunitinib: 4 weeks of sunitinib of 50 mg orally each day then 2 weeks of no medication until progression.
Arm/Group | Everolimus | Sunitinib
Number analyzed (Participants) | 57 | 51
Participants | 18 | 27

4. Secondary Outcome: Overall Survival of the First Line Therapy
Description: The amount of time each participant is alive from the start of the first line therapy.
Time Frame: 17 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus | Sunitinib
Number analyzed (Participants) | 35 | 33
months | 14.9 [8.0 to 23.4] | 16.2 [14.2 to NA] — insufficient number of participants with events

5. Secondary Outcome: Number of Participants With Best Overall Response for First Line Medication
Description: The best overall response for each participant was determined by using the Response Evaluation Criteria for Solid Tumors (RECIST). The responses are Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progression Disease (PD). CR is the disappearance of the cancer everywhere in the participant. PR is at least a 30 % reduction in the measured tumors from baseline. SD is no discernible change in the presence of cancer. Progressive disease is an increase of at least 20% of the measured cancer from the cancer's smallest measure.
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus | Sunitinib
Number analyzed (Participants) | 35 | 33
Participants
  Complete Response | 0 | 0
  Partial Response | 1 | 3
  Stable Disease | 26 | 21
  Progressive Disease | 8 | 9

ADVERSE EVENTS:
Time Frame: All Cause Mortality was measure for 8 Years. Adverse events and Serious adverse events were measured for 1 year.
Description: Adverse events that were related to either medication were documented and graded for severity according to the Common Terminology Criteria of Adverse Events (CTCAE) version 3. Grades increase in severity from 1 - 5. Grade 1 is a mild change. Grade 2 is a moderate change. Grade 3 is a sever change and may require hospitalization. Grade 4 is life threatening. Grade 5 is death.
Groups:
- Everolimus: 4 weeks of everolimus 10 mg orally each day then 2 weeks of no medication until progression.
- Sunitinib: 4 weeks of sunitinib 50 mg orally each day then 2 weeks of no medication until progression. At progression will crossover to everolimus.
Arm/Group | Everolimus | Sunitinib
All-Cause Mortality (participants affected / at risk) | 21/57 | 20/51
Serious Adverse Events (participants affected / at risk) | 12/57 | 14/51
Other Adverse Events (participants affected / at risk) | 38/57 | 46/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=57) | Sunitinib (N=51)
CNS cerebrovascular ischemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Platelets (Immune system disorders) | 0 (0) | 3 (3)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain (Nervous system disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyponatremia (Investigations) | 0 (0) | 2 (2)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=57) | Sunitinib (N=51)
Hypoalbuminenia (General disorders) | 3 (4) | 12 (23)
Alkaline phosphatase (Metabolism and nutrition disorders) | 5 (8) | 5 (6)
ALT (Metabolism and nutrition disorders) | 12 (15) | 17 (21)
Anorexia (Endocrine disorders) | 9 (13) | 8 (9)
AST (General disorders) | 19 (33) | 23 (30)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (6) | 7 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (6) | 13 (28)
Hypercholestremia (Metabolism and nutrition disorders) | 27 (48) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (14) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 3 (4)
Creatinine (Metabolism and nutrition disorders) | 20 (37) | 23 (50)
Diarrhea (Gastrointestinal disorders) | 17 (33) | 26 (131)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 (25) | 17 (34)
Edema (Respiratory, thoracic and mediastinal disorders) | 12 (25) | 18 (38)
Fatigue (General disorders) | 33 (96) | 46 (196)
Hyperglycemia (Metabolism and nutrition disorders) | 31 (74) | 17 (26)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 8 (10)
Dyspepsia (General disorders) | 2 (4) | 13 (17)
Anemia (Blood and lymphatic system disorders) | 33 (88) | 33 (100)
Hemoglobinuria (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 7 (9)
Hypertension (Endocrine disorders) | 2 (3) | 20 (33)
Infection (Infections and infestations) | 8 (9) | 4 (4)
Leukocytes (Blood and lymphatic system disorders) | 12 (26) | 30 (112)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (9)
Depression (Nervous system disorders) | 0 (0) | 3 (3)
Mucositis (Gastrointestinal disorders) | 36 (111) | 27 (72)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Nail changes (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (4)
Nausea (Gastrointestinal disorders) | 17 (31) | 29 (115)
Neuropathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (9)
Neutrophils (Nervous system disorders) | 3 (6) | 20 (79)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6) | 6 (11)
Pain (General disorders) | 14 (31) | 21 (44)
Platelets (Blood and lymphatic system disorders) | 11 (21) | 32 (79)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (4) | 6 (8)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 6 (11)
Proteinuria (Renal and urinary disorders) | 15 (37) | 16 (27)
Rash (Skin and subcutaneous tissue disorders) | 19 (52) | 24 (97)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 6 (18)
Hypernatremia (Metabolism and nutrition disorders) | 5 | 10
Dysgeusia (Nervous system disorders) | 6 (6) | 19 (20)
Hypothyroidism (Endocrine disorders) | 2 (2) | 3 (3)
Hypertriglyderidemia (General disorders) | 22 (45) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (10) | 12 (44)
Watery eye (Eye disorders) | 4 (6) | 2 (4)
Weight loss (Metabolism and nutrition disorders) | 5 (5) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 10 (11) | 8 (10)
Hypokalemia (Metabolism and nutrition disorders) | 5 (16) | 10 (17)
Proteinuria (Renal and urinary disorders) | 25 (47) | 22 (33)
Rash (Skin and subcutaneous tissue disorders) | 29 (64) | 21 (53)
Hyponatremia (Metabolism and nutrition disorders) | 5 (10) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 4 (4) | 11 (28)
Dysgeusia (Nervous system disorders) | 10 (10) | 25 (27)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 38 (78) | 2 (3)
Vomiting (Gastrointestinal disorders) | 11 (15) | 16 (50)
Watery eye (Eye disorders) | 9 (13) | 6 (16)
Weight loss (Metabolism and nutrition disorders) | 6 (6) | 2 (3)
UTI (Infections and infestations) | 4 (5) | 3 (3)
Magnesuim low (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 4 (4) | 7 (12)
Hand foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (3) | 22 (70)
Hypernatremia (Metabolism and nutrition disorders) | 8 (13) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/66/NCT01185366/Prot_SAP_000.pdf